CLINICAL TRIAL: NCT06385639
Title: A Double-blind, Randomized Clinical Study, Compared With Placebo to Assess the Efficacy and Safety of a Probiotic Product Containing Four Probiotic Strains to Support Digestive Environment and Homeostasis of Gut Microbiota
Brief Title: Efficacy and Safety of Probiotic Products for Digestive Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: WK2024005
Record Dates: First submitted 2024-04-22; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Healthy Adult
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic Group (Experimental): Two sachets/day probiotics, before breakfast and dinner, respecitvely
  Interventions: Dietary Supplement: Probiotic
- Placebo Group (Placebo Comparator): Maltodextrin, Two sachets/day probiotics, before breakfast and dinner, respecitvely
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — This clinical trial will last for 10 days, and each subject will have 4 follow-up visits (Day -1, Day 0, Day 10, Day 20).

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of the probiotic product as an everyday gut health product in supporting digestive environment and homeostasis of gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female subject age 18-60 years at screening
2. Healthy subject according to investigator judgement based on screening data
3. Subjects must be either of non-childbearing potential, or if of childbearing potential, they must be abstinent or have practiced adequate contraception for the entire study
4. Subjects who have not smoked in the past 1 month prior to screening
5. Subjects with a healthy and balanced diet, including adequate fiber intake in their food consumption
6. Subject or subject's legally acceptable representatives have the ability to comply with the trial protocol
7. Signed informed consent from the subjects or subject's legally acceptable representatives (must be obtained before any trial related activities)

Exclusion Criteria:

1. History of presence of diabetes, immunodeficiency disorders, or chronic illness
2. Regular use of medications known to affect the gastrointestinal system or alter gut microbiota composition, including but not limited to antibiotics, and immunosuppressants
3. Have continuous, daily use of probiotic or probiotic containing products within 1 month prior to randomization
4. Pregnant, planning a pregnancy or lactating female (urinary pregnancy test will be applied to female subjects at screening)
5. Change type of diet during study
6. Any known allergy or intolerance to any of the ingredients in the formulation of the product under study
7. History of drug, alcohol or other substance abuse, or other factors that limit their ability to cooperate during the study
8. History of or presence of eating disorder
9. Subject whose condition does not make them eligible to the study, according to the investigator

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-25 (Estimated); Primary Completion 2024-05-25 (Estimated); Study Completion 2024-06-25 (Estimated)

PRIMARY OUTCOMES:
Intestinal health | 10 days
  Changes in short-chain fatty acid (SCFA) from baseline to day 10

CONTACTS AND LOCATIONS:
Locations (1):
- Danang@Equilab-Int.Com, Jakarta, Pusat, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided